CLINICAL TRIAL: NCT00774618
Title: Prospective Trial of Operative Management of Rib Fracture Non-Union
Brief Title: Evaluation of Surgical Treatment on Pain and Disability for Chronic, Non-healing Rib Fracture
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: ACUTE Innovations, LLC (Industry)
Responsible Party: Principal Investigator, John C. Mayberry, Professor of Surgery, Oregon Health and Science University
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: IRB e4073
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Rib Fracture
Keywords: Rib Fracture; Thoracic Injuries; Flail Chest; Rib Fracture Repair; Rib Fracture ORIF; Chronic rib fractures; Non-healing rib fractures; Rib Fracture Non-union
MeSH Terms: conditions — Rib Fractures; Thoracic Injuries; Flail Chest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resection (Experimental): Those subjects undergoing resection with or without plate fixation
  Interventions: Device: Resection with or without plate fixation
- Nonoperative (No Intervention): These patients were not considered candidates for surgical intervention by the investigators, declined surgical intervention, or did not receive insurance approval for surgery

INTERVENTIONS:
Device: Resection with or without plate fixation — Some enrolled subjects will undergo rib fracture surgery at OHSU. Devices used in the repair of rib fracture non-union could include RibLoc® or BioBridge ™. RibLoc® is a U-shaped permanent device that secures to the rib with screws locking from the front to the back of the metal plate (through the rib). BioBridge ™ is a resorbable, non-permanent device that stabilizes the ribs. Both devices are designed to stabilize the rib fracture non-union and promote healing of the non-union rib. For some patients, it may be determined that resection of the rib fracture non-union without an implanted device is the most appropriate treatment. The goal of surgical intervention is to improve the pain and disability associated with rib fracture non-union in appropriate patients.
  Arms: Resection

SUMMARY:
Individuals with non-healing rib fractures may experience significant pain and disability. This is called rib fracture non-union, an unusual problem and one that most physicians have little experience with. The investigators hypothesize that surgical repair of rib fracture non-union is clinically efficacious and safe in 6 month follow-up. The objective of this study is to evaluate how repairing non-healing rib fractures affects pain and disability.

DETAILED DESCRIPTION:
Rib fractures are a painful and disabling injury commonly found among trauma patients. According to the National Center for Health Statistics, approximately 350,000 people with rib fractures were treated in emergency and ambulatory care departments in the United States in the year 2006. The Healthcare Cost and Utilization Project's Nationwide Inpatient Sample for the year 2003 indicated that 102,000 patients with rib fractures were admitted to U.S. hospitals, representing 7 % of all injured patients.

Within the past decade a subgroup of patients with symptomatic rib fracture non-unions has been identified. These are patients who present to primary care physicians and surgical clinics more than 3 months, or in some cases several years, following a rib fracture injury with complaints of rib pain associated with persistent fracture movement. They are usually told by their physician that surgical intervention is either unnecessary or fruitless and are treated with chronic pain management regimens. The true incidence and the long-term outcome of this syndrome are completely unknown.

At OHSU, the investigators have had a long interest in the indications for and the outcomes of rib fracture repair. One of the first of three nearly simultaneous reports of successful surgical intervention of symptomatic rib fracture non-union originated here at OHSU in 2001. Two other successful case reports have appeared more recently. The investigators are currently being contacted frequently by patients or their physicians, mostly out of state, for consideration of rib fracture non-union repair. Our ongoing experience with rib fracture non-union repair has been favorable, but the investigators believe that a prospective clinical study with at least 6 months of post-operative outcome is necessary. In addition, because the insurance company approval process for surgical intervention for rib fracture non-union is often 2 - 3 months and occasionally longer, the investigators have an opportunity to follow the intermediate-term natural history of rib fracture non-unions for several months prior to surgical intervention.

The rationale for conducting this study is to demonstrate in a prospective study that the RibLoc ® repair system is durable and safe in a population of patients with rib fracture non-union. Although this clinical outcome data is not required by the FDA to market and implant this prosthesis, the investigators believe that to establish the clinical benefit of the RibLoc ® device for non-union repair, prospectively collected outcome data are necessary. Investigators may use other FDA approved devices (i.e. BioBridge ™ Bioresorbable Bone Fracture Plate), or determine that no device is indicated (i.e. rib resection without hardware). The investigators expect to learn about clinical outcomes for surgical care in this group of patients, both with the use of a device, and without.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 18 years of age
2. Subjects must have rib fracture non-union (3 months or greater since injury), confirmed with Chest CT or MRI
3. The subject will have signed an IRB approved written informed consent and HIPAA authorization to participate in the study
4. Subjects will be able to participate in interviews with study staff and complete study surveys reliably

Exclusion Criteria:

1. Subjects who are enrolled in another investigational treatment trial
2. Subjects who have received an investigational drug or device within 30 days of enrollment
3. Female subjects who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-10; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of employment or disability status | At study entry (day 1) and 2 month intervals for up to 12 months.

SECONDARY OUTCOMES:
quality of life evaluation | At study entry (day 1) and 2 month intervals for up to 12 months.
  (Rand 36-Item Short Form Health Survey)
an assessment of rib fracture pain | At study entry (day 1) and 2 month intervals for up to 12 months.
  McGill Pain Questionnaire or MPQ
complications related to injury or treatment | At study entry (day 1) and 2 month intervals for up to 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: John C Mayberry, MD, FACS, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Cacchione RN, Richardson JD, Seligson D. Painful nonunion of multiple rib fractures managed by operative stabilization. J Trauma. 2000 Feb;48(2):319-21. doi: 10.1097/00005373-200002000-00023. No abstract available. PMID 10697096
- [Background] Ng AB, Giannoudis PV, Bismil Q, Hinsche AF, Smith RM. Operative stabilisation of painful non-united multiple rib fractures. Injury. 2001 Oct;32(8):637-9. doi: 10.1016/s0020-1383(01)00017-1. No abstract available. PMID 11587704
- [Background] Slater MS, Mayberry JC, Trunkey DD. Operative stabilization of a flail chest six years after injury. Ann Thorac Surg. 2001 Aug;72(2):600-1. doi: 10.1016/s0003-4975(00)02262-1. PMID 11515905
- [Background] Beelen R, Rumbaut J, De Geest R. Surgical stabilization of a rib fracture using an angle stable plate. J Trauma. 2007 Nov;63(5):1159-60. doi: 10.1097/01.ta.0000222536.91745.b4. No abstract available. PMID 17514061
- [Background] Richardson JD, Franklin GA, Heffley S, Seligson D. Operative fixation of chest wall fractures: an underused procedure? Am Surg. 2007 Jun;73(6):591-6; discussion 596-7. PMID 17658097
- [Background] Sales JR, Ellis TJ, Gillard J, Liu Q, Chen JC, Ham B, Mayberry JC. Biomechanical testing of a novel, minimally invasive rib fracture plating system. J Trauma. 2008 May;64(5):1270-4. doi: 10.1097/TA.0b013e31804a7fd5. PMID 18469649
- [Background] Nirula R, Diaz JJ Jr, Trunkey DD, Mayberry JC. Rib fracture repair: indications, technical issues, and future directions. World J Surg. 2009 Jan;33(1):14-22. doi: 10.1007/s00268-008-9770-y. PMID 18949513